CLINICAL TRIAL: NCT02999295
Title: A Multicenter, Phase 1/2 Study of Ramucirumab Plus Nivolumab as Second-line Therapy in Participants With Gastric or GEJ Cancer
Brief Title: A Phase 1/2 Study of Ramucirumab Plus Nivolumab in Participants With Gastric or GEJ Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Center, Japan (Other Government)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry); Fiverings Co., Ltd. (Other)
Responsible Party: Principal Investigator, Ken Kato, Head Physician, National Cancer Center, Japan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCH-1611
Record Dates: First submitted 2016-12-19; First posted 2016-12-21 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Gastric Cancer; Gastroesophageal Junction Region (GEJ) Cancer
MeSH Terms: conditions — Stomach Neoplasms; Neoplasms | interventions — Ramucirumab; Nivolumab

ARMS (2):
- Phase 1 (Experimental): Ramucirumab: 8 mg/kg, every two week Nivolumab: 3.0 mg/kg or 1.0 mg/kg (optional), every two weeks
  Interventions: Biological: Ramucirumab; Biological: Nivolumab
- Phase 2 (Experimental): Ramucirumab: 8 mg/kg, every two week Nivolumab: recommended dose established in the phase 1, every two weeks
  Interventions: Biological: Ramucirumab; Biological: Nivolumab

INTERVENTIONS:
Biological: Ramucirumab — Ramucirumab (8 mg/kg) is administered.
  Other Names: LY3009806
Biological: Nivolumab — Nivolumab (3.0 mg/kg or 1.0 mg/kg) is administered.
  Other Names: ONO-4538

SUMMARY:
The main purpose of this study is to evaluate the safety and efficacy of the combination therapy of ramucirumab and nivolumab in participants with advanced or recurrent unresectable gastric or GEJ cancer.

ELIGIBILITY:
Inclusion Criteria:

* Advanced or recurrent unresectable gastric or GEJ cancer
* Histologically confirmed adenocarcinoma (papillary adenocarcinoma, tubular adenocarcinoma or poorly differentiated adenocarcinoma), signet-ring cell carcinoma, mucinous adenocarcinoma or hepatoid adnocarcinoma
* Patients with normal oral intake
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Patients who have measurable target lesion
* Patients has a refractory or intolerant pretreatment by pyrimidine fluoride anticancer agent and platinum-based anticancer agent
* Patients with adequate organ function
* Patients with no pretreatment history including ramucirumab, nivolumab or other therapies targeting control of T cells
* Patients with written informed consent

Exclusion Criteria:

* Patients have double cancer
* Patients have infection required systemic therapy
* Known central vervous system (CNS) metastasis
* Patients with history of pneumonitis or pulmonary fibrosis
* Patients with history of serious anaphylaxis induced by antibody preparation
* Patients who have known active autoimmune disease or history of chronic recurrent autoimmune disease
* Female who is pregnant, lactating or suspected pregnancy
* Patients with psychosis or dementia to interfere to obtain informed consent appropriately

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicities (DLTs) | Phase 1, course 1 (up to 28 days)
  Number of participants with dose limiting toxicities (DLTs)
Progression free survival rate after 6 months | from baseline to 6 months
  Progression free survival rate after 6 months

SECONDARY OUTCOMES:
Number of participants with adverse events | from baseline to date of treatment cessation, approximately 24 months
  Number of participants with adverse events
Objective response rate (ORR) | from baseline to date of disease progression, approximately 24 months
  percentage of participants with with a best response of complete response (CR) or partial response (PR)
Disease control rate (DCR) | from baseline to date of disease progression, approximately 24 months
  percentage of participants with with a best response of CR, PR or stable disease (SD)
Overall survival (OS) | from baseline to date of death, approximately 24 months
  Overall survival (OS)
Progression free survival (PFS) | from baseline to date of disease progression or death, approximately 24 months
  Progression free survival (PFS)

CONTACTS AND LOCATIONS:
Overall Officials: Ken Kato, M.D. / Ph.D., Principal Investigator — Department of Gastrointestinal Medical Oncology, National cancer center hospital
Locations (1):
- National Cancer Center Hospital, Tokyo, Japan